CLINICAL TRIAL: NCT00727025
Title: Closing Linear Incisions in Plastic Surgery: A Randomized Clinical Trial Comparing a New Coaptive Film Device Versus Standard Subcuticular Sutures for Scar Quality, Patient Comfort, and Closure Time
Brief Title: Randomized Controlled Trial of Subcuticular Skin Closure Versus Steri-strip S Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPHS 20069
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2013-05

CONDITIONS: Breast Hypertrophy; Abdominal Elastosis; Breast Reconstruction
Keywords: skin closure devices; linear scars
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: wound closure device (Steri-Strip™) — wound closure with steri-strip S
  Other Names: 3M™ Steri-Strip™ S Surgical Skin Closure

SUMMARY:
Purpose: The aims of this randomized clinical trial are:

1. to assess scar quality from the patient and surgeon perspectives
2. to assess patient comfort in the days immediately following surgery
3. to assess the time taken to complete closure in the operating room.
4. the financial benefit or cost for the institution of using Steri Strip S will also be estimated.

Two closure methods will be compared, a new coaptive film device (Steri Strip S) versus standard subcuticular sutures. The linear incisions will include the standard incision segments utilized for an inverted-T closure for bilateral breast reduction and the transabdominal incision segments utilized for abdominoplasty or TRAM flap harvest.

Our hypothesis is that incisions segments closed with Steri Strip S compared to standard subcuticular closure, will yield scars of better cosmetic quality, in shorter time to closure, with novice and expert surgeons, for both bilateral breast reduction and abdominoplasty surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for enrollment if they agree to provide informed consent, are at least 18 years of age, in generally good health, and available for follow-up in the 5-7 month time frame.

Exclusion Criteria:

* Women known to be pregnant, minors, patients potentially incompetent to provide informed consent or complete the surveys described in our protocol will be excluded from this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Kerrigan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Kerrigan CL, Homa K. Evaluation of a new wound closure device for linear surgical incisions: 3M Steri-Strip S Surgical Skin Closure versus subcuticular closure. Plast Reconstr Surg. 2010 Jan;125(1):186-194. doi: 10.1097/PRS.0b013e3181c2a492. PMID 20048611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all woman undergoing bilateral breast reduction using the Wise pattern approach. Pts were recruited between Feb 2006 and Sept 2007
Pre-assignment Details: Patients declined
Groups:
- All Participants: Participants randomized to have one segment of wounds closed with steri-strip device and the other wound segment closed with traditional suture closure.
Period: Overall Study
Arm/Group | All Participants
Started | 74
Completed | 51
Not Completed | 23
Not completed — Physician Decision | 23

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 74
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Scar Quality at 6 Months Postoperative
Description: Patients used a rating scale with range of 1-9 with 1 being the best scar and 9 being the worst scar. Patients had photos of scars within this range to anchor their choices.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Wounds Closed With Device: segment of wounds closed with steri-strip device
- Wounds Closed With Suture: wound segments closed with traditional suture
Arm/Group | Wounds Closed With Device | Wounds Closed With Suture
Number analyzed (Participants) | 51 | 51
units on a scale | 3.8 (2.9) | 2.6 (2.1)

2. Secondary Outcome: Patient Postoperative Incisional Comfort
Description: Using a comfort scale from 0-10 with 0 being very uncomfortable and 10 being very comfortable
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wounds Closed With Device | Wounds Closed With Suture
Number analyzed (Participants) | 51 | 51
units on a scale | 5.8 (2.7) | 6.9 (2.0)

3. Primary Outcome: Time to Perform Wound Closure
Description: Time from completion of deep dermal closure to complete closure of wound, either by steri-strip application or by subcuticular suture
Time Frame: intraoperatively
Population: those who completed application of devices intraoperatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Steri-strip Closure | Suture Closure
Number analyzed (Participants) | 51 | 51
minutes | 2.0 (1.1) | 4.6 (1.6)

ADVERSE EVENTS:
Arm/Group | Wounds Closed With Device | Wounds Closed With Suture
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

LIMITATIONS AND CAVEATS:
1. patients not blinded
2. surgeons rated photographs of scars, while the patients were rating their actual scars.
3. All patients were caucasian

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No